CLINICAL TRIAL: NCT04778267
Title: The Effectiveness of Combined U.S. Guided Erector Spinae and Pecto-intercostal Fascial Plane Blocks Versus U.S.Guided Thoracic Paravertebral Block in Controlling Perioperative Pain in Modified Radical Mastectomy, a Blinded Randomized Controlled Trial
Brief Title: Effectiveness of Combined Erector Spinae and Pecto-intercostal Fascial Plane Blocks Versus Thoracic Paravertebral Block in Perioperative Pain in Modified Radical Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Sara Farouk Kassem Habib, principal investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-342-2020
Record Dates: First submitted 2021-02-15; First posted 2021-03-03 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Modified Radical Mastectomy
MeSH Terms: interventions — Bupivacaine; dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: The effectiveness of combined ultrasound guided erector spinae and pectointercostal fascial plane blocks versus ultrasound guided thoracic paravertebral block in controlling perioperative pain in modified radical mastectomy, a blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: randomization table created by a researcher who is not involved in the study. The researcher will assign the random ID to each patient and a blinded anesthesiologist will use this ID while collecting the postoperative data in the surgical ward. The block interventions of this study will be done by the same anesthesiologist (well trained to use US-guided regional techniques) while pre-operative and postoperative data collection will be done by another anesthesiologist blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPVB (thoracic paravertebral block) (Active Comparator): TPVB will be performed in the sitting position A high frequency linear ultrasound probe will be applied in the parasagittal plane approximately 2-3 cm lateral to the midline till identification of the 3rd thoracic vertebra (T3) in the same side of surgery. Then the transducer will be moved progressively more medially until transverse processes are identified.The image acquired will have the transverse process located superiorly and an image of lower rib located inferiorly on the screen.The needle tip is to be observed to enter through the superior costotransverse ligament and loss of resistance sensation will be experienced. After confirming the anterior displacement of pleura with 2-3 mL of local anesthetic (LA), 30 ml of 0.25% bupivacaine and 4 mg dexamethasone will be administered for the block.
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Dexamethasone phosphate
- ES-PI (erector spinae-pectointercostal block) (Experimental): ESPB In the second group (ES-PI) Using a high frequency linear ultrasound probe, it will be located in a longitudinal orientation at the level of T3 spinous process and then will be placed 3 cm laterally from the midline to the side involved in the surgery. .a 22-gauge block needle will be inserted in-plane at an angle of 30-40°. 20 mL of 0.25% bupivacaine hydrochloride and 3 mg dexamethasone will be injected in the plane deeper to the erector spinae muscle.
  PIPB While the patient is in the supine position, a high frequency linear probe will be placed parallel to the long axis of the sternum at a distance 2-3 cm from the attachment of the second rib and sternum to identify the Pectoralis major muscle, external intercostal muscles and the second rib in the superficial plane. by separation of fascial layers of between the external intercostal and the pectoralis muscles, a total of 10 ml of 0.25% bupivacaine and 1 mg dexamethasone will be injected.
  Interventions: Drug: Bupivacaine Hydrochloride; Drug: Dexamethasone phosphate

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — We hypothesize that combined ESPB and PIPB are as effective as TPVB in controlling perioperative pain in patients undergoing modified radical mastectomy (MRM) with lesser complications using bupivacaine hydrocloride
  Other Names: marcaine
Drug: Dexamethasone phosphate — used as additive to bupivacaine
  Other Names: decadrone

SUMMARY:
Erector spinae plane block (ESPB) is a new evolving fascial pain block in the era of regional anaesthesia. ESPB was applied in varieties of surgeries and provided an eminent role in trauma patient especially those with fracture ribs. ESPB exhibits simple, safe and easy technique with minimal or no sympathetic blockade effects, thus gaining popularity in wide range of surgeries. The optimum effective dose of local anaesthetic, the effective volume of drug used for desired dermatomes. Comparison with different regional blocks is preferable to know the optimum analgesic technique for those population of patients (4). Many studies have already compared solo ESPB with thoracic epidural analgesia (TEA), thoracic paravertebral block (TPVB), serratus anterior plane block (SAPB) and pectoral nerves block. Only few case reports described the combination effect of rhomboid intercostal, transversus thoracic muscle and parasternal plane blocks to ESPB in modified radical mastectomy.

DETAILED DESCRIPTION:
patients scheduled for modified radical mastectomy and axillary dissection under general anesthesia (GA) will be included in the study. The patients will be randomly allocated by a computer-generated table into one of the two study groups.Thoracic paravertebral block group (TPV group) and combined erector spinae and pecto-intercostal fascial plane blocks group (ES-PI group).

0.25% bupivacaine and 1 mg dexamethasone will be injected with different volumes in each block.

The first time to ask for rescue analgesia post-operatively will be measured. Using MedCalc Software version 14 (MedCalc Software bvba, Ostend, Belgium), 24 patients (12 patients per group) were calculated for a relative difference of 10% (0.635 hours) in the time to first analgesic request between both groups, with a study power of 95% and an alpha error of 0.05. This number will be increased to 30 patients (15 patients per group) to compensate for possible dropouts.

Analysis of data will be performed using the Statistical Package for Social Science (SPSS) software, version 21 for Microsoft Windows (SPSS Inc., Chicago, iL, USA). Categorical data will be reported as numbers and percentages and will be analyzed using the chi-squared test. Continuous data will be checked for normality using the Kolmogorov-Smirnov test. Normally distributed data will be presented as means (standard deviations) and will be analyzed using the unpaired student t-test. Skewed data will be expressed as medians(quartiles) and will be analyzed using the Mann Whitney U test. For repeated measures, a two-way repeated measures ANOVA will be used to evaluate block (between-groups factor) and time (repeated measures)". Post-hoc pairwise comparison will be performed using the Bonferroni test. A P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* • 18-60 years of age

  * ASA I-II
  * Elective unilateral modified radical mastectomy with axillary lymph node dissection
  * Body weight (50-90 kg)

Exclusion Criteria:

* • Patient refusal

  * Known allergy to any of the study drugs
  * Bleeding disorders (platelets < 50 000, PC <60%, INR>1.5)
  * Infection at the site of needle puncture or sepsis
  * Obesity (BMI > 30 kg/m2)
  * Chronic opioid user eg; morphine addict
  * Chronic pain disease eg certain cancer patients, rheumatological disease
  * Inability to comprehend or use the numeric rating pain scoring system
  * Psychiatric illness eg, psychiatric patients on hypnotic treatment

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
The first time to ask for rescue analgesia post-operatively | 48 hours
  after how many hours postoperatively the patient will ask for analgesia

SECONDARY OUTCOMES:
The total postoperative opioid consumption (in the first 48 hrs) | 48 hours
  total milligrams of opioid given to the patient in the 48 hours postoperatively
NRS scores | 48 hours postoperative
  Postoperative pain will be assessed, using numeric rating scale (NRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Kase Al Aini teaching hospital, Cairo, Kasr Al Aini, Egypt

IPD SHARING:
Plan to Share IPD: No